CLINICAL TRIAL: NCT00346619
Title: Investigating the Time of Nelfinavir Treatment Necessary for an Increase in Thymic Naive T Cells in Adults.
Brief Title: Determining the Amount of Time Needed for Nelfinavir to Boost the Immune System in Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1298-05
Record Dates: First submitted 2006-06-28; First posted 2006-06-30 (Estimated); Last update posted 2010-01-20 (Estimated); Status verified 2010-01

CONDITIONS: Immune Response
MeSH Terms: interventions — Nelfinavir

INTERVENTIONS:
Drug: Nelfinavir

SUMMARY:
Our group has shown that HAART increases the thymic production of naïve T cells in the healthy adult, thereby boosting the immune system. We propose to investigate the amount of and length of Nelfinavir therapy necessary to increase those cells in adults. Subjects will be treated with Nelfinavir, and blood will be sampled at variable times to determine the immune response in peripheral blood.

DETAILED DESCRIPTION:
Blood will be collected at several time points during the study. DNA will be isolated from peripheral blood lymphocytes (PBL) and assessed for signal point (sj) TREC content relative to genomic CCR5 copies by real time PCR in a spectoflourometic thermal cycler. TREC values will be expressed as TREC copy number per copies of CCR5 or TREC/PBLs.

We anticipate that we will confirm our previous observations that nelfinavir therapy will increase TRECs, indicating naive T cell production from the thymus. The proposed study will determine the time course of the anticipated increase in TREC/PBLs.

ELIGIBILITY:
Healthy individuals between the ages of 20 and 100. Exclusion criteria include the following: HIV, HBV/HCV positive, known sensitivity to protease inhibitors, oral intake contraindicated, diabetes mellitus diagnosed within the last six months, and any of the following medications: cisapride, amiodarone, terfenadine, rifampin/rifabutin, phenobarbital, pinozide, St. John's wort, ergot derivatives, quinidine, astemazole, carbemazapine, phenytoin, midazolam, triazolam, and simvastatin.

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2005-10; Primary Completion 2007-10 (Actual); Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
Will confirm that HIV protease inhibitors increase thymic naïve T-cell production and determine the dose and time needed to increase thymic T-cell production in adults.

CONTACTS AND LOCATIONS:
Overall Officials: Stacey R. Vlahakis, M.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

REFERENCES:
- [Derived] Rizza SR, Tangalos EG, McClees MD, Strausbauch MA, Targonski PV, McKean DJ, Wettstein PJ, Badley AD. Nelfinavir monotherapy increases naive T-cell numbers in HIV-negative healthy young adults. Front Biosci. 2008 Jan 1;13:1605-9. doi: 10.2741/2784. PMID 17981652